CLINICAL TRIAL: NCT05551702
Title: Treating Depression With Text Delivered Counseling (Depression Study 2.0)
Brief Title: Treating Depression With Text Messaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Michael Mason, Principal Investigator, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dep 2.0
Record Dates: First submitted 2022-09-13; First posted 2022-09-23 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-05

CONDITIONS: Moderate Depression
Keywords: Cognitive Behavioral Therapy; Text-Based Intervention

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the treatment group or the waitlist control group. The treatment group will receive 8 weeks of the text based intervention (CBT-txt) and complete surveys at baseline, 1 month, 2 months and 3 months. The waitlist control group will only do surveys at baseline, 1 month, 2 months, and 3 months and will then have the option of receiving the intervention after their 3 months of study participation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): This arm will receive 8 weeks of the text-based intervention (CBT-txt). CBT-txt is a version of Cognitive Behavioral Therapy tailored to be delivered by automated text message. This arm will also complete surveys at baseline, 1 month, 2 months, and 3 months.
  Interventions: Behavioral: CBT-txt
- Waitlist Control (No Intervention): This arm will not receive the text-based intervention during study participation. These participants will only complete surveys at baseline, 1 month, 2 months, and 3 months and will be given the option to receive CBT-txt after they complete study participation.

INTERVENTIONS:
Behavioral: CBT-txt — Cognitive Behavioral Therapy delivered via automated text messaging.
  Arms: Treatment

SUMMARY:
The purpose of the research study is to investigate whether CBT-txt, a counseling program delivered by text messages is effective in stopping or reducing depressive symptoms. CBT-txt is based on a counseling program that has been proven to reduce depression when delivered in-person and on the web, but has not yet been tested or shown to be effective when delivered by text.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, participants will complete online screening assessments. Once eligibility is confirmed, participants will be randomized either to the intervention group or to the waitlist-control group. Those who are randomized to the intervention group will receive the 8-week text intervention via smartphone and complete assessments at baseline, 1 month, 2 months, and 3 months. Those who are randomized to the waitlist-control group will only complete the assessments at baseline, 1 month, 2 months, and 3 months. Participants who are initially assigned to the waitlist-control group can choose to receive the text intervention once their 3-month participation is complete.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 25 years old
* a score of at least 5 on the PHQ-9 (indicating elevated depression symptoms

Exclusion Criteria:

* treatment for depression during the past three months
* endorse suicide ideation on the PHQ-9*
* lack of access to a text-capable phone
* unable or unwilling to commit to two months of follow-up
* not fluent in English.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Beck Depression Inventory II at 2 Months | Baseline, 1 Month, 2 Month, 3 Month
  A 21-item instrument for measuring the severity of depression in adults and adolescents aged 13 years and older. Minimum score =0, Maximum=63. Higher scores indicate more depression.
Change from Baseline Beck Depression Inventory II at 3 Months | Baseline, 1 Month, 2 Month, 3 Month
  A 21-item instrument for measuring the severity of depression in adults and adolescents aged 13 years and older. Minimum score =0, Maximum=63. Higher scores indicate more depression.

SECONDARY OUTCOMES:
Change from Baseline Types of Thinking Cognitive Distortion Scale at 2 Months | Baseline, 1 Month, 2 Months, 3 Months
  A 10 item scale using scenarios to help recognize cognitive distortions. Minimum score = 20, Maximum = 140. Higher scores equal more cognitive distortions.
Change from Baseline Types of Thinking Cognitive Distortion Scale at 3 Months | Baseline, 1 Month, 2 Months, 3 Months
  A 10 item scale using scenarios to help recognize cognitive distortions. Minimum score = 20, Maximum = 140. Higher scores equal more cognitive distortions.
Change from Baseline Perseverative Thinking Questionnaire at 2 Months | Baseline, 1 Month, 2 Months, 3 Months
  A 15 item scale rating statements about negative experiences or problems to identify repetitive negative thinking. Minimum score = 0, Max 60. Higher scores equal more perseverative thinking.
Change from Baseline Perseverative Thinking Questionnaire at 3 Months | Baseline, 1 Month, 2 Months, 3 Months
  A 15 item scale rating statements about negative experiences or problems to identify repetitive negative thinking. Minimum score = 0, Max 60. Higher scores equal more perseverative thinking.
Change from Baseline Behavioral Activation for Depression Scale at 2 Months | Baseline, 1 Month, 2 Months, 3 Months
  A 9 items scale to measure how and when participants become activated during behavioral activation treatment. Minimum score = 0, Max = 54. Higher scores equal more behavioral activation.
Change from Baseline Behavioral Activation for Depression Scale at 3 Months | Baseline, 1 Month, 2 Months, 3 Months
  A 9 items scale to measure how and when participants become activated during behavioral activation treatment. Minimum score = 0, Max = 54. Higher scores equal more behavioral activation.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Mason, PhD, Principal Investigator — University of Tennessee-Knoxville
Locations (1):
- University of Tennessee-Knoxville, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mason MJ, Coatsworth JD, Zaharakis N, Russell M, Brown A, McKinstry S. Testing Mechanisms of Change for Text Message-Delivered Cognitive Behavioral Therapy: Randomized Clinical Trial for Young Adult Depression. JMIR Mhealth Uhealth. 2023 Jul 11;11:e45186. doi: 10.2196/45186. PMID 37432723